CLINICAL TRIAL: NCT04585542
Title: Comparison of Potassium Binders in the ER
Acronym: KBindER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Wei Ling Lau, Associate Professor in Nephrology, Dpt of Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS# 2020-5780
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Hyperkalemia; Oral Potassium Binders
Keywords: Emergency Department
MeSH Terms: conditions — Emergencies | interventions — polyethylene glycol 3350; polystyrene sulfonic acid; patiromer; sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and ER physicians are blinded to study drug allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Polyethylene glycol 3350 (MiraLax) (Experimental): Participants will be randomized to one of four study arms. They will receive one dose of the study drug.
  One study arm is the nonspecific laxative MiraLax (one dose of 17g). Since constipation can contribute to hyperkalemia, this arm will study the effect of treating constipation instead of direct cation exchange for potassium in the gut.
  Interventions: Drug: Polyethylene Glycol 3350
- Sodium polystyrene sulfonate (Kayexalate) (Experimental): Participants will be randomized to one of four study arms. They will receive one dose of the study drug.
  The potassium binder drugs of interest include sodium polystyrene sulfonate (one dose of 30g), patiromer (one dose of 25.2g), and sodium zirconium cyclosilicate (one dose of 15g).
  Interventions: Drug: Sodium Polystyrene Sulfonate Oral Suspension [SPS]
- Patiromer (Veltassa) (Experimental): Participants will be randomized to one of four study arms. They will receive one dose of the study drug.
  The potassium binder drugs of interest include sodium polystyrene sulfonate (one dose of 30g), patiromer (one dose of 25.2g), and sodium zirconium cyclosilicate (one dose of 15g).
  Interventions: Drug: Patiromer
- Sodium zirconium cyclosilicate (Lokelma) (Experimental): Participants will be randomized to one of four study arms. They will receive one dose of the study drug.
  The potassium binder drugs of interest include sodium polystyrene sulfonate (one dose of 30g), patiromer (one dose of 25.2g), and sodium zirconium cyclosilicate (one dose of 15g).
  Interventions: Drug: Sodium zirconium cyclosilicate

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — Nonspecific laxative comparison group.
  Other Names: MiraLax
  Arms: Polyethylene glycol 3350 (MiraLax)
Drug: Sodium Polystyrene Sulfonate Oral Suspension [SPS] — Potassium binder to treat hyperkalemia.
  Other Names: Kayexalate
  Arms: Sodium polystyrene sulfonate (Kayexalate)
Drug: Patiromer — Potassium binder to treat hyperkalemia.
  Other Names: Veltassa
  Arms: Patiromer (Veltassa)
Drug: Sodium zirconium cyclosilicate — Potassium binder to treat hyperkalemia.
  Other Names: Lokelma
  Arms: Sodium zirconium cyclosilicate (Lokelma)

SUMMARY:
Compare efficacy of 3 oral potassium binders (cation exchange resins) on lowering blood potassium, in hospital patients with acute hyperkalemia.

DETAILED DESCRIPTION:
Adult patients presenting to the Emergency Room or currently hospitalized at UC Irvine (not in ICU level of care) with plasma potassium >5.5 mEq/L (who meet inclusion/exclusion criteria and provide written informed consent) will be randomized to a one-time dose of one of the following oral medications:

1. Sodium polystyrene sulfate (SPS)
2. Patiromer (Veltassa)
3. Sodium zirconium cyclosilicate (Lokelma)
4. Nonspecific laxative: polyethylene glycol 3350 (MiraLax)

Participants will receive standard-of-care hyperkalemia therapy as well.

Blood potassium will be checked at 2 and 4 hours after dose of study drug. Participants will complete a symptom and palatability questionnaire at 4 hours.

The purpose of this research study is to determine the effects of various potassium binders (SPS, patiromer, zirconium) vs a non-specific laxative (MiraLax) in hospital patients found to have elevated blood potassium > 5.5 mEq/L. Hyperkalemia is a fairly common electrolyte disorder with varying levels of severity. Moderate hyperkalemia is in the range 5.5-5.9 mEq/L while severe hyperkalemia is ≥6.0 mEq/L or if patient is symptomatic: muscle weakness/paralysis or with EKG changes (e.g., peaked T waves, widening QRS, arrhythmias including ventricular fibrillation or asystole). Hyperkalemia is most commonly associated with kidney insufficiency, metabolic acidosis, and the use of medications such as renin-angiotensin-aldosterone system inhibitors.

In an emergency, the main goal is to reverse adverse cardiac effects and shift potassium into cells using interventions such as insulin/glucose and albuterol. However, these are only temporary measures. To remove potassium from the body, agents or interventions that may be used include cation exchange resins (potassium binders), loop diuretics, or dialysis. For over 50 years the only available oral cation exchange resin has been sodium polystyrene sulfonate. In recent years, two new agents (patiromer and zirconium) have been approved by the FDA for chronic management of hyperkalemia.

The cation exchange resins have not been studied head-to-head for acute hyperkalemia. This is a critical knowledge gap since acute hyperkalemia poses a significant burden on the healthcare system. In claims data analysis of 80,000 patients, half with hyperkalemia and half without, the patients with hyperkalemia had 4 times higher rate of inpatient admissions, 7 times longer average length of stay, and 30-day hospital readmission rate 14.21% vs 9.86% in the non-hyperkalemia cohort. The findings from our study will help inform decision-making guidelines for the treatment of acute hyperkalemia.

ELIGIBILITY:
Inclusion Criteria:

* Plasma potassium > 5.5 mEq/L
* Age ≥18 years
* Patient able to provide written informed consent

Exclusion Criteria:

* Recent bowel surgery
* Ileus or bowel obstruction
* Pseudohyperkalemia signs and symptoms, such as excessive fist clenching, hemolyzed blood specimen, severe leukocytosis or thrombocytosis
* Pregnancy
* Active psychiatric disorder
* Diabetic ketoacidosis or hyperkalemia caused by any condition for which a therapy directed against the underlying cause of hyperkalemia would be a better treatment option
* Dialysis session expected within 4 hours after randomization
* History of hypersensitivity to sodium polystyrene sulfonate resin or patiromer
* Concurrent use of sorbitol (due to increased risk of intestinal necrosis when used with sodium polystyrene sulfonate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in blood potassium level | Plasma potassium level measured at 2 and 4 hours after study drug was administered
  The investigators will compare the change in blood potassium after administration of the study drug, in the acute setting.

SECONDARY OUTCOMES:
Length of ER or hospital stay | Up to 60 days after study drug was administered
  The investigators will compare length of ER or hospital stay associated with each study drug, obtained from medical chart review.
Change in calcium, phosphorus and magnesium | Measured at 2 and 4 hours after study drug was administered
  The investigators will compare the effect of each study drug on blood calcium, phosphorus and magnesium levels, in the acute setting.
Dialysis yes/no within 8 hours | Within 8 hours of study drug being administered
  The investigators will assess whether dialysis was needed to manage hyperkalemia, and whether dialysis requirement was affected by the study drug given. This will be assessed from medical chart review.
Palatability and side effects (patient subjective rating) | 4 hours after study drug was administered
  Participants will complete a 1-page brief survey assessing for potential study drug side effects including bloating, nausea, diarrhea and palpitations (answers are yes/no). Participants will also rate the palatability of the study drug using a 1-5 scale, with 5 being the best score (most palatable and easy to swallow).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. De-identified dataset can be made available to other researchers, please contact PI Dr. Lau.

REFERENCES:
- [Background] Leon SJ, Harasemiw O, Tangri N. New therapies for hyperkalemia. Curr Opin Nephrol Hypertens. 2019 May;28(3):238-244. doi: 10.1097/MNH.0000000000000500. PMID 30865167
- [Background] Betts KA, Woolley JM, Mu F, Xiang C, Tang W, Wu EQ. The Cost of Hyperkalemia in the United States. Kidney Int Rep. 2017 Nov 14;3(2):385-393. doi: 10.1016/j.ekir.2017.11.003. eCollection 2018 Mar. PMID 29725642
- [Derived] Canas AE, Troutt HR, Jiang L, Tonthat S, Darwish O, Ferrey A, Lotfipour S, Kalantar-Zadeh K, Hanna R, Lau WL. A randomized study to compare oral potassium binders in the treatment of acute hyperkalemia. BMC Nephrol. 2023 Apr 5;24(1):89. doi: 10.1186/s12882-023-03145-x. PMID 37016309